CLINICAL TRIAL: NCT06398886
Title: Effects of Ericksonian Hypnotherapy Versus Cognitive Behavioral Therapy on Prolonged Grief Among University Students in Istanbul: A Randomized Controlled Trial
Brief Title: Ericksonian Hypnosis Versus CBT for Prolonged Grief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Metin Çınaroğlu, Asistant Professor, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nisantasi-Hypnosis
Record Dates: First submitted 2024-04-18; First posted 2024-05-03 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Prolonged Grief Symptoms
Keywords: Prolonged Grief; Ericksonian Hypnosis; Cognitive Behavioral Therapy; Randomized Controlled Trial
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: There have been 3 groups, CBT, Hypnosis and Waiting, each group has 13 participants, CBT and Hypnosis group has taken 8 sessions each and waiting list group took none.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ericksonian Hypnosis Group (Experimental): Ericksonian hypnotherapy provided an alternative approach, with 8 sessions designed to harness the power of indirect suggestion, metaphors, and personal storytelling to navigate the complexities of prolonged grief. Early sessions focused on establishing a therapeutic alliance and utilizing personal strengths and inner resources. Techniques such as guided imagery were used to facilitate a healthy connection with the symptoms, fostering a sense of peace and acceptance. Subsequent sessions aimed to reframe the loss, integrating it into the individual's life narrative in a way that honored the past while promoting openness to future possibilities. This approach sought to cultivate a sense of personal growth and resilience, emphasizing the individual's capacity to find meaning and continue moving forward.
  Interventions: Behavioral: Ericksonian Hypnosis; Behavioral: Cognitive Behavioral Therapy
- Waiting List (Control) (Active Comparator): No intervention has been provided for this group.
  Interventions: Behavioral: Ericksonian Hypnosis; Behavioral: Cognitive Behavioral Therapy
- Cognitive Behavioral Therapy (Experimental): The Cognitive Behavioral Therapy (CBT) intervention for prolonged grief was carefully structured into an 8-session manualized program, tailored to address the multifaceted nature of grief among university students. Initially, participants were introduced to the CBT model of grief, focusing on understanding the relationship between thoughts, feelings, and behaviors in the context of their loss. Key components included identifying and challenging maladaptive thoughts related to the loss, employing gradual exposure to avoided situations, and developing coping strategies for managing intense emotions and fostering resilience. Special emphasis was placed on rebuilding meaningful life activities and social connections, acknowledging the loss while encouraging engagement with life's ongoing demands.
  Interventions: Behavioral: Ericksonian Hypnosis; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Ericksonian Hypnosis — The Ericksonian hypnosis intervention was designed to create a nurturing and therapeutic setting, specifically tailored to the unique challenges of prolonged grief faced by university students. This approach focused on accessing the subconscious, using symbolic and imaginative techniques to facilitate change. The goal was to alleviate the emotional pain associated with prolonged grief and to empower students to adapt more effectively to their loss. This intervention highlighted the transformative potential of Ericksonian methods in addressing deep-seated emotional issues through gentle and indirect therapeutic modalities.
Behavioral: Cognitive Behavioral Therapy — The CBT intervention aimed to provide a supportive and healing environment, addressing the specific challenges of prolonged grief within a university student population. The focus was on developing concrete skills to manage the cognitive and behavioral aspects of grief. This approach sought to mitigate the pain of prolonged grief and empower students to adapt more healthily to their loss, emphasizing practical strategies for change and coping. Participants were encouraged to actively engage in exercises that challenged their thought patterns and promoted behavioral adjustments tailored to their individual needs.

SUMMARY:
Effects of Ericksonian Hypnotherapy Versus Cognitive Behavioral Therapy on Prolonged Grief Among University Students in Istanbul: A Randomized None-clinical Controlled Trial

This randomized controlled trial explores the efficacy of Ericksonian Hypnotherapy versus Cognitive Behavioral Therapy (CBT) in mitigating symptoms of prolonged grief among university students in Istanbul. With a backdrop of transitional academic and socio-emotional challenges, 39 students who experienced significant loss and exhibited symptoms of prolonged grief were enrolled. Participants were randomly assigned to undergo Ericksonian Hypnotherapy, CBT, or placed on a waiting list (control group), each with 13 individuals. The study uniquely positions itself in Istanbul, leveraging the city's cultural context to examine grief processing in an urban, academically engaged population. Utilizing the Prolonged Grief Scale, Beck Depression Inventory, and SCL-90 Symptom Checklist for assessment, the interventions were evaluated for their effectiveness in reducing grief and associated psychological symptoms.

DETAILED DESCRIPTION:
Background Grief is a universal, deeply personal response to loss. While most individuals eventually adjust, some experience prolonged grief disorder (PGD), marked by intense longing, preoccupation with the deceased, and difficulty engaging with life, significantly impacting well-being.

The transition to university is a critical developmental period for young adults, often accompanied by new challenges and, at times, loss. University students, navigating adulthood away from traditional support systems, may experience grief more profoundly, affecting their academic performance, relationships, and mental health. Despite its importance, grief among university students remains underexplored.

Istanbul, with its diverse cultural landscape and large student population, provides a unique context to study prolonged grief. The city's dynamic environment and academic pressures may shape students' grief experiences, influenced by cultural attitudes toward loss and mourning.

This study investigates the effectiveness of Ericksonian hypnotherapy and CBT in treating prolonged grief among university students in Istanbul, addressing a critical gap in grief interventions for young adults and contributing to mental health support within academic settings.

Rationale Prolonged grief disorder is a persistent form of bereavement, distinct from normal grief and major depression, that significantly impairs functioning. CBT, with its structured approach to modifying maladaptive thoughts and behaviors, is effective in treating various psychological disorders, including prolonged grief. Despite its benefits, not all individuals respond to CBT, underscoring the need for alternative therapies.

Ericksonian hypnotherapy, developed by Milton H. Erickson, uses indirect suggestion, metaphors, and storytelling to facilitate change, emphasizing individual inner resources and the unconscious mind. Its personalized, experiential nature aligns well with university students' developmental stage and cognitive flexibility. The symbolic methods may also resonate within Istanbul's culturally rich context, offering a potentially sensitive approach to grief therapy.

Comparing Ericksonian hypnotherapy to CBT for prolonged grief is essential due to their differing therapeutic mechanisms, the lack of research in university settings, and the potential to expand grief intervention options. This study addresses a critical gap by evaluating these therapies among Istanbul's university students, aiming to enhance psychological well-being and academic success.

Objectives

The primary aim of this randomized non-clinical controlled trial is to evaluate and compare the effectiveness of Ericksonian hypnotherapy and CBT in addressing symptoms of prolonged grief among university students in Istanbul. This comparison seeks to achieve several key objectives:

1. Assess the Reduction in Prolonged Grief Symptoms: To quantitatively measure and compare the reduction in symptoms of prolonged grief among participants, as evaluated by the Prolonged Grief Scale, following the completion of Ericksonian hypnotherapy and CBT interventions. This objective seeks to identify which therapeutic approach is more effective in alleviating the core symptoms of prolonged grief.
2. Evaluate Changes in Associated Psychological Symptoms: To examine and compare the impact of Ericksonian hypnotherapy and CBT on associated psychological symptoms, including depression and overall psychological distress, as measured by the Beck Depression Inventory and Prolonged Grief Scale, respectively. This objective aims to understand the broader psychological benefits of each therapy in treating prolonged grief.
3. Investigate Participant Engagement and Satisfaction: To assess and compare participant engagement and satisfaction with Ericksonian hypnotherapy versus CBT, incorporating participant feedback and session attendance rates. This objective is important for evaluating the acceptability and feasibility of both therapeutic approaches among university students.
4. Explore Cultural and Contextual Factors: To explore how cultural and contextual factors inherent to the student population in Istanbul may influence the effectiveness and reception of Ericksonian hypnotherapy and CBT for prolonged grief. This objective recognizes the importance of cultural sensitivity in psychological interventions and aims to provide insights into tailoring therapies to specific populations.

Methodology Study Design This research employed a randomized controlled trial design to evaluate the effectiveness of Ericksonian hypnotherapy versus CBT in treating prolonged grief among university students in Istanbul. The study aimed to recruit 150 volunteers who had experienced loss and exhibited symptoms of grief. To ensure participants did not present with other significant psychological symptoms that could confound the results, the SCL-90 Symptom Checklist was utilized alongside the Prolonged Grief Scale and the Beck Depression Inventory.

Participants Participants were university students in Istanbul who volunteered for the study, meeting the inclusion criteria of having experienced a significant loss and showing symptoms of prolonged grief as assessed by the Prolonged Grief Scale. Exclusion criteria included undergoing psychotherapy during the past year, significant psychological disorders as identified by the SCL-90, and inability to commit to the full duration of the study. After initial screening, 39 participants who scored high on the Prolonged Grief Scale were selected and randomly assigned into three groups: Ericksonian hypnotherapy, CBT, and a waiting list control, with 13 participants in each group.

Interventions The Cognitive Behavioral Therapy (CBT) intervention for prolonged grief was carefully structured into an 8-session manualized program, tailored to address the multifaceted nature of grief among university students. Initially, participants were introduced to the CBT model of grief, focusing on understanding the relationship between thoughts, feelings, and behaviors in the context of their loss. Key components included identifying and challenging maladaptive thoughts related to the loss, employing gradual exposure to avoided situations, and developing coping strategies for managing intense emotions and fostering resilience. Special emphasis was placed on rebuilding meaningful life activities and social connections, acknowledging the loss while encouraging engagement with life's ongoing demands.

Ericksonian hypnotherapy provided an alternative approach, with 8 sessions designed to harness the power of indirect suggestion, metaphors, and personal storytelling to navigate the complexities of prolonged grief. Early sessions focused on establishing a therapeutic alliance and utilizing personal strengths and inner resources. Techniques such as guided imagery were used to facilitate a healthy connection with the symptoms, fostering a sense of peace and acceptance. Subsequent sessions aimed to reframe the loss, integrating it into the individual's life narrative in a way that honored the past while promoting openness to future possibilities. This approach sought to cultivate a sense of personal growth and resilience, emphasizing the individual's capacity to find meaning and continue moving forward.

Both interventions aimed to provide a supportive and healing environment, addressing the specific challenges of prolonged grief within a university student population. The CBT group worked on concrete skills for tackling the cognitive and behavioral aspects of their grief, while the Ericksonian group delved into the subconscious to elicit change through more symbolic and imaginative processes. Despite their methodological differences, both therapies shared the goal of mitigating the pain of prolonged grief and empowering students to adapt more healthily to their loss. Participants in the waiting list control group were offered information on available grief counseling resources upon conclusion of the study, ensuring they too had access to support.

Data Collection and Measures Data were collected at three time points: before the start of the sessions, after the fourth session, and immediately after the eighth and final session. The Prolonged Grief Scale and Beck Depression Inventory were administered at each time point to assess changes in grief intensity, depressive symptoms, and overall psychological distress, respectively.

Measurement Tools Prolonged Grief Scale (PGS): The Prolonged Grief Scale is a specialized instrument designed to assess the symptoms and severity of prolonged grief disorder (PGD) among individuals. This scale consists of items that measure the core symptoms of PGD, including persistent yearning for the deceased, difficulty accepting the death, a sense of disbelief regarding the loss, and marked emotional pain related to the bereavement. Each item is rated on a Likert scale, allowing for a quantifiable measure of grief intensity. The reliability and validity of the PGS have been established in various populations, making it a robust tool for identifying individuals suffering from PGD (Prigerson et al., 2021).

Beck Depression Inventory (BDI): The Beck Depression Inventory is a widely used 21-item self-report inventory measuring the severity of depression in adolescents and adults. Each item corresponds to a specific symptom or attitude related to depression, such as sadness, pessimism, feelings of failure, and dissatisfaction with life. Respondents are asked to rate how they have felt over the past two weeks on a four-point scale ranging from 0 to 3, with higher scores indicating more severe depressive symptoms. The BDI's reliability and validity are well-documented, making it a valuable tool for assessing depressive symptoms in conjunction with grief (Beck et al., 1987).

SCL-90 Symptom Checklist: The SCL-90 is a 90-item self-report symptom inventory designed to reflect the psychological symptom patterns of community, medical, and psychiatric respondents. It measures nine primary symptom dimensions, including depression, anxiety, hostility, and paranoid ideation, and provides an overall index of distress, the Global Severity Index (GSI). Each item is rated on a five-point scale of distress, from "not at all" to "extremely." This tool allows for the comprehensive assessment of a range of psychological symptoms and distress levels, ensuring that participants do not have significant comorbid psychological conditions that could influence the study's outcomes (Derogatis & Unger, 2010).

Data Collection Process Recruitment and Screening: Potential participants were recruited through university networks and advertisements, targeting students who had experienced a significant loss. Interested volunteers underwent a preliminary screening using a SCL-90 to confirm eligibility based on the study's inclusion and exclusion criteria. This included assessing their grief experience, previous therapy, and any psychological disorders.

Baseline Assessment: Eligible participants completed the Prolonged Grief Scale and Beck Depression Inventory as part of the baseline assessment. These tools were administered in a controlled environment to ensure confidentiality and reduce potential biases. The baseline data collection aimed to establish initial levels of grief, depression, and psychological distress among participants, serving as a reference point for subsequent analyses.

Randomization and Group Assignment: Following baseline assessment, participants were randomly assigned to one of three groups: Ericksonian hypnotherapy, CBT, or waiting list control. Randomization was performed using a computer-generated sequence to ensure equal distribution of participants across the groups and minimize selection bias.

Intervention and Follow-up Assessments: Participants in the Ericksonian hypnotherapy and CBT groups attended 8 sessions of their respective therapies. Data were collected again after the fourth session and immediately after the eighth session using the same measurement tools (PGS, BDI). This repeated measurement allowed for the tracking of changes in grief and depression over the course of the interventions.

Data Handling and Analysis: All collected data were coded and entered into a secure database for analysis. Participant confidentiality was maintained throughout the study, with personal identifiers removed or anonymized. Data analysis focused on comparing pre- and post-intervention scores within and between groups, assessing the effectiveness of Ericksonian hypnotherapy and CBT in reducing symptoms of prolonged grief and associated psychological distress.

Statistical Analysis Data analysis was performed using SPSS software. Descriptive statistics were employed to characterize the sample demographics and baseline measures. The primary analysis involved comparing the pre- and post-intervention scores within and between the treatment and control groups using repeated measures ANOVA, followed by post hoc comparisons to identify specific differences. Effect sizes were calculated to determine the magnitude of the interventions' impacts. Significance levels were set at p < 0.05 for all tests.

Ethical Considerations The study was approved by the Institutional Review Board (IRB) of İstanbul Nişantaşı University No: 2023/2, ensuring that it met ethical standards for research involving human participants. Informed consent was obtained from all participants, emphasizing the voluntary nature of participation, the confidentiality of their responses, and their right to withdraw from the study at any time without penalty.

ELIGIBILITY:
Inclusion Criteria

* Age Range: Participants must be aged between 18 and 35 years.
* Loss Experience: Participants should have experienced the loss of someone significant.
* Grief Intensity: Participants must score 25 or above on the Prolonged Grief Scale (PG-13).
* Psychological Health: Participants should not exhibit other psychopathological symptoms, apart from those associated with grief, as measured by the Symptom Checklist-90 (SCL-90).
* Commitment to Participation: Participants must be able and willing to attend all 8 full sessions.

Exclusion Criteria

* Age Limitations: Individuals under 18 or older than 35 years are excluded.
* Psychiatric Health: Individuals with any psychiatric diagnosis or those who have been on psychiatric medication within the last year are excluded.
* Availability: Individuals who cannot commit to attending all 8 sessions are excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Metin Çınaroğlu, phd, Study Chair — Assistant Professor in Psychology department; Eda Yılmazer, phd, Study Director — Assistant Professor in Psychology Department; Fadime Çınar, phd, Principal Investigator — Associated Professor and head of faculty of health sciences
Locations (1):
- Metin Çınaroğlu, Arnavutköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 university students were recruited through campus advertisements and social media, targeting individuals who had experienced significant loss and exhibited symptoms of prolonged grief. Interested students completed an initial online screening, which included the Symptom Checklist-90 and a sociodemographic form. Of these, 39 met the inclusion criteria, while 111 were excluded due to factors such as ongoing psychological treatment, major psychiatric conditions, or scheduling conflicts.
Period: Overall Study
Arm/Group | Ericksonian Hypnosis Group | Waiting List (Control) | Cognitive Behavioral Therapy
Started | 13 | 13 | 13
Completed | 13 | 13 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 150 university students were recruited; 39 met eligibility criteria and were randomized into Ericksonian Hypnotherapy (EH), Cognitive Behavioral Therapy (CBT), or a waitlist control group (13 per group). Both EH and CBT participants completed 8 sessions, with no dropouts. Grief and depression scales were administered at baseline, midpoint, and post-intervention. All participants completed the study, ensuring full data for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ericksonian Hypnosis Group | Waiting List (Control) | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 13 | 39
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.04 (0.15) | 21.0 (0.17) | 20.8 (0.18) | 21.03 (0.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 29
  Male | 4 | 3 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 7 | 9 | 11 | 27
  Iran | 2 | 2 | 0 | 4
  Egypt | 1 | 1 | 0 | 2
  Azerbaijan | 2 | 1 | 0 | 3
  Uzbekistan | 1 | 0 | 1 | 2
  Iraq | 0 | 0 | 1 | 1
Baseline PGS Scores [Mean (Standard Deviation); unit: Points] — The Prolonged Grief Scale (PGS) was used to measure the intensity of grief-related symptoms at baseline. Scores range from [X] to [Y], with higher scores indicating greater grief intensity.
  Points | 34 (7) | 21 (10) | 24 (7) | 26.33 (8.43)

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Grief Scale
Description: The Prolonged Grief Scale (PGS) was used to measure the intensity of grief-related symptoms at baseline. The PGS consists of 13 items rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (overwhelmingly). Total scores range from 0 to 52, with higher scores indicating greater intensity of prolonged grief symptoms. This scale has demonstrated reliability and validity in assessing grief severity among diverse populations Number of Items: The scale consists of 13 items. Scoring for Each Item: Each item is rated on a 5-point scale, ranging from 0 (not at all) to 4 (overwhelmingly).
  Minimum Score: The minimum possible score on the PG-13 is 0, indicating no symptoms of prolonged grief.
  Maximum Score: The maximum possible score is 52, indicating severe symptoms of prolonged grief.
Time Frame: Data were collected at baseline, midpoint (4 weeks), and post-intervention (8 weeks
Population: All 39 participants completed the study. Data analysis was performed using the Prolonged Grief Scale scores collected at baseline, midpoint, and post-intervention
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Ericksonian Hypnosis Group | Waiting List (Control) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 13 | 13 | 13
points
  Baseline | 34 (7) | 21 (10) | 24 (7)
  Midpoint | 26 (11.55) | 19 (8.49) | 18 (10.77)
  Post-Intervention | 13 (11.55) | 17 (8.49) | 12 (10.77)

2. Primary Outcome: Beck Depression Inventory
Description: Number of Items: The BDI-II consists of 21 items. Scoring for Each Item: Each item has a set of four statements that are scored on a scale from 0 to 3, reflecting increasing severity of a specific symptom.
  Minimum Score: The minimum possible score on the BDI-II is 0, which would indicate no reported symptoms of depression.
  Maximum Score: The maximum possible score is 63, reflecting severe depression.
  The total score is interpreted as follows:
  0-13: Minimal depression 14-19: Mild depression 20-28: Moderate depression 29-63: Severe depression
Time Frame: 8 weeks
Population: All 39 participants completed the study. BDI-II scores were collected at baseline, midpoint (4 weeks), and post-intervention (8 weeks) from all participants.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Ericksonian Hypnosis Group | Waiting List (Control) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 13 | 13 | 13
points
  Baseline | 38.15 (11.22) | 25.54 (12.31) | 21.38 (8.89)
  4 weeks | 33 (9.93) | 24.62 (11.83) | 16.77 (6.58)
  8 weeks | 26.08 (9.82) | 25.69 (12.34) | 13.23 (6.31)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 12-week period, spanning from the initiation of the first therapy session to the post-treatment follow-up assessment. This timeframe ensured comprehensive monitoring of any potential adverse events throughout the study duration
Description: Adverse events, including all-cause mortality, were systematically monitored throughout the 12-week study period. Participants self-reported during therapy sessions and follow-ups. No adverse events, including all-cause mortality, were observed in any group. All 39 participants (13 per group) completed the study without reporting adverse events.
Arm/Group | Waiting List (Control) | Cognitive Behavioral Therapy | Ericksonian Hypnosis Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT06398886/Prot_SAP_000.pdf